CLINICAL TRIAL: NCT03408613
Title: Obstructive Sleep Apnea and Glucose Metabolism
Acronym: OSAGM
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: equipment recall
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Bettina Mittendorfer, Senior Associate Dean for Research, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201710015
Record Dates: First submitted 2017-12-01; First posted 2018-01-24 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Sleep Apnea; Glucose Metabolism Disorders
Keywords: Obstructive Sleep Apnea; Glucose Metabolism
MeSH Terms: conditions — Sleep Apnea Syndromes; Glucose Metabolism Disorders; Sleep Apnea, Obstructive | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Positive Airway Pressure (PAP) (Experimental): A registered polysomnographic technologist will perform a titration starting at 4 cm water (H2O) and adjust this value as needed to identify the optimal pressure to achieve an Apnea Hypopnea Index (AHI) <5 (including rapid eye movement sleep in the supine position). After PAP titration, subjects will be instructed to use the machine at the optimal pressure every night for 3 months. Compliance will be defined as: ≥4 hours use on 70% of nights and average use ≥6 hours per night.
  Interventions: Procedure: Positive Airway Pressure
- Supplemental Oxygen (O2) (Experimental): Subjects randomized to night-time supplemental oxygen will complete an overnight oxygen titration protocol in the clinical research unit. Initially, subjects will receive 0.5 liters oxygen (O2)/min; the delivery rate will then be increased by 0.5 l/min until oxygen saturation (SaO2) is ≥88%. The optimal O2 delivery rate determined during this study will be used for the intervention. The oxygen concentrators used at home will record cumulative hours of use to provide an objective measure of adherence (monitored weekly). Compliance will be defined as ≥6 h average use per night..
  Interventions: Procedure: Supplemental Oxygen
- Sham (Sham Comparator): Subjects in the sham treatment group will complete the oxygen titration protocol described for the night-time supplemental oxygen group, except that their oxygen concentrator will have been covertly modified to deliver room air at a rate of 0.5 l/min.
  Interventions: Procedure: Sham
- Controls (No Intervention): Subjects without OSA will be recruited and complete all testing for primary outcome measures, but will not undergo any intervention.

INTERVENTIONS:
Procedure: Positive Airway Pressure — See arm/group description
  Arms: Positive Airway Pressure (PAP)
Procedure: Supplemental Oxygen — See arm/group description
  Arms: Supplemental Oxygen (O2)
Procedure: Sham — See arm/group description
  Arms: Sham

SUMMARY:
Many adults who are overweight have obstructive sleep apnea (OSA) which disrupts sleep and makes it difficult to breath during the night. OSA increases the risk for a person to become insulin resistant and diabetic. It is not known why OSA causes this problem, i.e., whether it is disrupted sleep or lack of oxygen., which can change how the body handles glucose in adipose tissue, muscle tissue and liver.

The purpose of this research study is to determine the key issues and mechanisms responsible for dysregulated glucose metabolism in people with OSA. The investigators will do this by comparing glucose metabolism in people who have OSA, and those who do not, and by evaluating the effect of treating OSA by providing continuous positive airway pressure (CPAP) or simply oxygen during the night.

The proposed study will evaluate the primary causes(s) (hypoxia, sleep fragmentation, or both) and pathophysiological mechanisms responsible for the OSA-associated metabolic abnormalities. Knowing the primary cause of Obstructive Sleep Apnea and pathophysiological mechanisms responsible for the OSA-associated metabolic abnormalities could help develop potentially novel therapeutic strategies to provide treatment for adults in improving OSA and associated comorbidities.

ELIGIBILITY:
General Inclusion Criteria (for all subjects):

* Age: ≥30 and ≤70 years,
* BMI: ≥30 and ≤45 kg/m2 or body fat ≥ 30 % for women and ≥ 25 % for men,
* Maximum body circumference <170 cm
* Weight stable (≤2% change)
* Untrained (≤1 h of structured exercise/wk) for at least 3 months before entering the study
* No diabetes (fasting blood glucose <126 mg/dl, 2h oral glucose tolerance test (OGTT) glucose <200 mg/dl, HbA1c ≤6.5%)

Sleep-related inclusion criteria:

Subjects without OSA:

* AHI <5/h of sleep;
* Oxygen desaturation index <3/h
* No known sleep disorders and periodic limb movement arousal index <15/h during polysomnography
* Reported sleep duration ≥6 h per night
* Regular sleep schedules (i.e. bedtime between 8 pm and 12 am and wake-time between 4 am and 8 am on all days of the week)

Subjects with OSA

* AHI ≥10/h of sleep (i.e., moderate to severe OSA)
* Oxygen desaturation index ≥4/h;
* No polysomnogram finding that would trigger immediate PAP treatment as per standard operating protocol in our sleep medicine center (a single SaO2 <50%, SaO2 <70% for >2 minutes, electrocardiogram pause >5 sec, or ventricular tachycardia >30 sec), because of the risk of a potentially adverse outcome if they are not randomized to the PAP group
* Periodic limb movement arousal index <15/h during polysomnography,
* Reported sleep duration ≥6 h per night,
* Regular night-time sleep schedules, defined as bedtime between 8 pm and 12 am and wake-time between 4 am and 8 am on all days of the week.

General Exclusion Criteria (for all subjects):

* Current treatment for previously diagnosed OSA;
* Self-reported severe difficulty sleeping in unfamiliar environments;
* Metal implants that are incompatible with magnetic resonance imaging;
* Controlled substances, tobacco products, dietary supplements, or medications known or suspected to affect sleep, breathing, upper airway muscle physiology, or glucose metabolism
* Evidence of disease (e.g., diabetes, congestive heart failure; chronic obstructive pulmonary disease; hypoventilation, defined as daytime partial pressure of carbon dioxide (pCO2) >45 mm Hg; major neurological or neuromuscular disorders; cancer; uncontrolled hypertension; etc.);
* Contraindications to supplemental oxygen or PAP (e.g., recent trans-sphenoidal surgery).
* Unwillingness or inability to provide informed consent
* Study physician considers subject to be unable to safely complete the study protocol

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-01-17 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Insulin mediated glucose disposal | 3 months
  The hyperinsulinemic-euglycemic clamp technique combined with isotope-labelled tracer infusions will be used to assess insulin mediated glucose rate of disappearance before and after treatment of OSA with three months of night-time supplemental oxygen, PAP, or sham.

SECONDARY OUTCOMES:
β-cell function | 3 months
  β-cell responsivity to glucose and the disposition index will be determined to characterize the insulin secretory response to glucose infusion and the relationship between insulin secretion and insulin sensitivity. This outcome will be determined by using an insulin-modified intravenous glucose tolerance test in conjunction with mathematical modelling and insulin sensitivity data from the hyperinsulinemic clamp.
Tissue oxygenation | 3 months
  Adipose and muscle tissue oxygenation, expressed as mmHg, will be evaluated in situ during the hyperinsulinemic-euglycemic clamp studies.
Body composition analysis | 3 months
  Detailed body composition analysis using dual energy x-ray absorptiometry (DXA) will provide the researchers with total and appendicular lean body and fat mass, expressed in grams of participants.

CONTACTS AND LOCATIONS:
Overall Officials: Bettina Mittendorfer, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cao C, Koh HE, Van Vliet S, Patterson BW, Reeds DN, Laforest R, Gropler RJ, Mittendorfer B. Increased plasma fatty acid clearance, not fatty acid concentration, is associated with muscle insulin resistance in people with obesity. Metabolism. 2022 Jul;132:155216. doi: 10.1016/j.metabol.2022.155216. Epub 2022 May 13. PMID 35577100
- [Derived] van Vliet S, Koh HE, Patterson BW, Yoshino M, LaForest R, Gropler RJ, Klein S, Mittendorfer B. Obesity Is Associated With Increased Basal and Postprandial beta-Cell Insulin Secretion Even in the Absence of Insulin Resistance. Diabetes. 2020 Oct;69(10):2112-2119. doi: 10.2337/db20-0377. Epub 2020 Jul 10. PMID 32651241